CLINICAL TRIAL: NCT01894464
Title: The Early Truancy Prevention Project
Acronym: ETPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A0207
Record Dates: First submitted 2013-06-27; First posted 2013-07-10 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Excessive Absenteeism by Primary School Students
Keywords: truancy; attendance; education; primary school; elementary school

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teacher led intervention (Experimental): Teachers will conduct teacher-led interventions that are individualized for each student to prevent emerging truancy among elementary students.
  Interventions: Behavioral: Teacher led intervention
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Teacher led intervention
  Arms: Teacher led intervention

SUMMARY:
The Early Truancy Prevention Project is designed to prevent elementary school truancy through teacher-led interventions that are individualized to meet student needs.

DETAILED DESCRIPTION:
The Early Truancy Prevention Project is an innovative intervention program designed to prevent elementary school truancy and later school dropout. The intervention model emphasizes the important role of teachers as change agents to address early attendance problems and emerging truancy. Specifically, the goals of this pilot project are: 1) to facilitate positive, trusting, and collaborative home-school relations and to promote a positive teacher-child relationship; 2) to provide teachers with timely information about a student's attendance pattern; and 3) to train and supervise teachers in the implementation of individualized attendance interventions to improve student attendance and prevent emerging truancy among elementary school students. As this is a pilot study, another important goal is to obtain teacher and administrator feedback to improve and refine all aspects of the project.

ELIGIBILITY:
Inclusion Criteria:

* all first and second grade teachers in 6 schools

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Percent of students who are truant | June, 2014
  Truancy is defined as 10 days absent during the academic year (approximately 10 months: August, 2013-June, 2014).

SECONDARY OUTCOMES:
Average number of absences per classroom | June, 2014
  Average number of absences per classroom during the academic year (approximately 10 months: August, 2013-June, 2014).

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Cook, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States